CLINICAL TRIAL: NCT00078169
Title: Motivational Enhancement for Spanish Speaking Individuals
Brief Title: Motivational Enhancement for Spanish Speaking Individuals - 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: University of Miami (Other)
Responsible Party: Kathleen Carroll, Ph.D., Yale University School of Medicine
Organization: National Institute on Drug Abuse (NIDA) (NIH)
Purpose: Treatment
Other Study IDs: NIDA-CTN-0021-1
Record Dates: First submitted 2004-02-19; First posted 2004-02-23 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-10

CONDITIONS: Substance-Related Disorders
Keywords: behavioral intervention
MeSH Terms: conditions — Substance-Related Disorders | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Behavior Therapy

SUMMARY:
The purpose of this study is to compare a three-session Spanish version of Motivational Enhancement Therapy (MET) to standard treatment to see how well MET engages and retains Spanish-speaking clients in outpatient substance abuse treatment.

ELIGIBILITY:
Inclusion Criteria:

All subjects included unless medical/psychiatrically unstable

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 463
Dates: Start 2003-11; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Treatment retention, drug and alcohol abstinence

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Carroll, Ph.D., Principal Investigator — Yale University
Locations (7):
- United States (7):
  - Island Grove RTC, Greeley, Colorado
  - Miami Behavioral Health, Miami, Florida
  - Counseling & Psychotherapy Institute, Albuquerque, New Mexico
  - The Life Link, Santa Fe, New Mexico
  - Narco Freedom (Bridge Plaza), Long Island City, New York
  - Changepoint - Cedar Hills Blvd, Portland, Oregon
  - Changepoint, Inc., Portland, Oregon